CLINICAL TRIAL: NCT00595179
Title: Intraoperative Assessment of Renal Perfusion Using Infrared Imaging
Brief Title: Intraperative Assessment of Renal Perfusion Using Infrared Imaging
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908042; 08-DK-N042
Record Dates: First submitted 2008-01-03; First posted 2008-01-16 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Transplantation
Keywords: Infrared; Imaging Techniques; Kidney Reperfusion; Pneumoperitoneum; Nephrectomy
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Current assessment of organ tissue viability by surgeons in the operating room is limited to crude estimates such as overt physical examination, measurement of laboratory values and physical measurements of vascular flow and resistance. The ability to non-invasively measure tissue perfusion and oxygenation would provide the surgeon an improved means to assess if an injured organ will survive. The recent development of real time infrared (IR) and Near Infrared Imaging Spectroscopy (NIRIS) digital cameras has allowed for the determination of tissue perfusion and oxygenation in a non-invasive fashion. Although in the early stages of development, the application of infrared and NIRS technology holds great promise to permit the surgeon to better assess the viability of tissues in ways that have not been possible. We propose to evaluate infrared and NIRS technology in the assessment of kidney allografts using data previously collected during recipient operations at the NIH.

DETAILED DESCRIPTION:
Current assessment of organ tissue viability by surgeons in the operating room is limited to crude estimates such as overt physical examination, measurement of laboratory values and physical measurements of vascular flow and resistance. The ability to non-invasively measure tissue perfusion and oxygenation would provide the surgeon an improved means to assess if an injured organ will survive. The recent development of real time infrared (IR) and Near Infrared Imaging Spectroscopy (NIRIS) digital cameras has allowed for the determination of tissue perfusion and oxygenation in a non-invasive fashion. Although in the early stages of development, the application of infrared and NIRS technology holds great promise to permit the surgeon to better assess the viability of tissues in ways that have not been possible. We propose to evaluate infrared and NIRS technology in the assessment of kidney allografts using data previously collected during recipient operations at the NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

NIH Transplant Reccipients of living related, living unrelated, and cadaveric kidney transplants who underwent intra-operative IR/NIRS imaging.

EXCLUSION CRITERIA:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-12; Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Disorders (NIDDK), 9000, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gorbach AM, Heiss J, Kufta C, Sato S, Fedio P, Kammerer WA, Solomon J, Oldfield EH. Intraoperative infrared functional imaging of human brain. Ann Neurol. 2003 Sep;54(3):297-309. doi: 10.1002/ana.10646. PMID 12953262